CLINICAL TRIAL: NCT02357602
Title: Dose Proportionality of TFV-DP in Mucosal Tissue, and Endogenous Nucleotide Quantification, After a Single Dose of GS-7340 in Women
Brief Title: Dose Proportionality of TFV-DP After a Single Dose of GS-7340 in Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 14-2797
Record Dates: First submitted 2015-01-14; First posted 2015-02-06 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Healthy
Keywords: Participants; HIV-1 negative
MeSH Terms: interventions — tenofovir alafenamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1. GS-7340 25mg (Experimental): The first 8 women on study will be assigned to take a single dose of 25mg TAF (1 tablet) orally.
  Interventions: Drug: GS-7340
- 2. GS-7340 10mg (Experimental): The 2nd group of 8 women will be sequentially assigned to take a single dose of 10mg TAF (1 tablet) orally.
  Interventions: Drug: GS-7340
- 3. GS-7340 5mg (Experimental): The final 8 women on study will be sequentially assigned to take a single dose of 5mg TAF (1/2 tablet) orally.
  Interventions: Drug: GS-7340

INTERVENTIONS:
Drug: GS-7340 — Medication is supplied in 10 or 25mg tablets, so subjects will receive either 1/2 or one tablet in a single dose.
  Other Names: TAF; Tenofovir Alafenamide

SUMMARY:
Purpose:

The purpose of this study is to characterize the dose-proportionality in the distribution of tenofovir alafenamide (TAF) and tenofovir (TFV) in plasma and mucosal tissues, and TFV-diphosphate (TFV-DP) in peripheral blood mononuclear cells (PBMCs) and mucosal tissues of healthy female subjects following a single oral dose of GS-7430 at 5mg, 10mg, and 25mg.

DETAILED DESCRIPTION:
Participants:

This study will consist of approximately 24 premenopausal healthy volunteer women between 18-49 years of age with an intact cervix, uterus, and gastrointestinal tract. Women will be enrolled in the study within 42 days of screening depending on the timing of their menstrual cycle in comparison to the screening visit, and then will be on study for 14 days, with follow-up 1-14 days after the end of study sampling. All study visits will be conducted in the North Carolina Translational and Clinical Sciences (NCTraCS) Clinical Translational Research Center (CTRC) at the University of North Carolina at Chapel Hill.

Procedures (methods):This is a Phase 1, single center, open-label, dose-ranging pharmacokinetic study of TFV and TFV-DP mucosal tissue concentrations measured after a single dose of GS-7340. Each arm is divided into three dosing groups: 5, 10, or 25mg. Participants will take a single dose of study drug within 7-14 days following the end of the subjects' menstrual period. Participants will be sequentially assigned to one of the three TAF doses and four biopsy schedules. Two women from each of the dosing groups will be assigned to one of four biopsy schedules for a total of 8 women per dosing group. Samples of blood plasma, cervicovaginal fluid (CVF), cervical tissue, vaginal tissue, and rectal tissue will be collected from participants at varying time points over the 14 days post-dose. Subjects will return to clinic within 14 days after the last sampling to complete a follow-up safety visit.

ELIGIBILITY:
Inclusion Criteria

1. Healthy pre-menopausal female subjects between the ages of 18 and 49 years, inclusive on the date of screening, with an intact gastrointestinal tract, uterus, and cervix.
2. All subjects must have an estimated calculated creatinine clearance (eCcr) of at least 80 mL/min
3. All subjects must have negative pregnancy tests, and be using an acceptable form of birth control
4. Body Mass Index (BMI) of approximately 18 to 34 kg/m²; and a total body weight > 45 kg (99 lbs).
5. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the trial.
6. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures.
7. Subject must have documentation of a normal pap smear within 36 months of the screening visit, no procedures for abnormal cervical/vaginal pathology in the last six months, at least one prior gynecological visit as part of subject's routine medical history.
8. Subject must be willing to abstain from sexual intercourse, douching, and all intravaginal and intrarectal objects and products for at least 72 hours prior to Day 1 until study completion.
9. Subject must be HIV-1 and Hepatitis B surface antigen negative
10. Subject must not be actively involved in the conception process.
11. Subject must be able to swallow pills and have no allergies to any component of the study products

Exclusion Criteria

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including documented drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
2. Subjects with a history of hysterectomy
3. Subjects who are pregnant, possibly pregnant or lactating
4. Subjects with a presence of vaginal discharge or genital bleeding at screening
5. History of febrile illness within five days prior to first dose.
6. Any condition possibly affecting drug absorption (eg, gastrectomy).
7. A positive urine drug screen.
8. A positive result for HIV, Hepatitis B or C
9. An untreated-positive test for syphilis, gonorrhea, Chlamydia, or trichomonas at screening, or symptomatic bacterial vaginosis.
10. Any laboratory chemistry or hematology result Grade 2 or greater according to the Division of Acquired Immunodeficiency Syndrome (DAIDS) Laboratory Grading Tables
11. Treatment with an investigational drug within 4 months preceding the first dose of trial medication.
12. History of regular alcohol consumption exceeding study limits
13. Participation in a clinical trial involving vaginal or rectal biopsies within 6 months preceding the first dose of trial medication.
14. Use of prescription or nonprescription drugs, vitamins, and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of trial medication and unable to avoid use during the study period until after the last sample is collected.
15. Blood donation of approximately 1 pint (500 mL) within 56 days prior to dosing.
16. History of sensitivity to heparin or heparin-induced thrombocytopenia.
17. Allergy to lidocaine or Monsel's solution.
18. Allergy to latex.
19. Abnormal pap smear in the past 36 months
20. Any degree of ectopy or abnormality evident during the pelvic exam at screening.
21. Any condition which, in the opinion of the investigator, is likely to interfere with follow-up or ability to take the study medication appropriately.
22. Unwilling or unable to comply with the dietary and concomitant drug restrictions in regard to study drug administration as outlined in the study procedures and prohibited medications sections.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-03; Primary Completion 2015-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Plasma Dose-Proportionality | Pre-dose and 1, 3, 6, 12, 24 hours, and 3, 7, 10, and 14 days following single dose
  To characterize the dose-proportionality in the distribution of TAF and TFV in the plasma of healthy female subjects following a single oral dose of GS-7340 at 5mg, 10mg, and 25mg. This will be used to develop a predictive pharmacokinetic model for TAF which will allow for TFVdp exposure predictions given a specific dose and dosing interval.
Tissue Dose-Proportionality | At 3, 6, 12 and 24 hours and 3, 7, 10 and 14 days following single dose
  To characterize the dose-proportionality in the distribution of TAF and TFV in mucosal tissues, and TFV-DP in mucosal tissues of healthy female subjects following a single oral dose of GS-7340 at 5mg, 10mg, and 25mg. This will be used to develop a predictive pharmacokinetic model for TAF which will allow for TFVdp exposure predictions given a specific dose and dosing interval.
PBMC Dose-Proportionality | Pre-dose and 3, 6, 12, 24 hours and 3, 7, 10, and 14 days following single dose
  To characterize the dose-proportionality in the distribution of TFV-DP in PBMCs of healthy female subjects following a single oral dose of GS-7340 at 5mg, 10mg, and 25mg. This will be used to develop a predictive pharmacokinetic model for TAF which will allow for TFVdp exposure predictions given a specific dose and dosing interval.

SECONDARY OUTCOMES:
Intra-subject variability in intracellular deoxyadenosine triphosphate (dATP) in peripheral blood | Pre-dose and 3, 6, 12, 24 hours and 3, 7, 10, and 14 days following single dose
  To determine intra-subject variability in intracellular dATP in PBMCs and ratios of TFVdp:dATP.
Inter-subject variability in intracellular deoxyadenosine triphosphate (dATP) in peripheral blood | Pre-dose and 3, 6, 12, 24 hours and 3, 7, 10, and 14 days following single dose
  To determine inter-subject variability in intracellular dATP in PBMCs and ratios of TFVdp:dATP.
Intra-subject variability in intracellular deoxyadenosine triphosphate (dATP) in mucosal tissues | At 3, 6, 12 and 24 hours and 3, 7, 10 and 14 days following single dose
  To determine intra-subject variability in intracellular dATP in cervical, vaginal, and rectal tissues and ratios of TFVdp:dATP.
Inter-subject variability in intracellular deoxyadenosine triphosphate (dATP) in mucosal tissues | At 3, 6, 12 and 24 hours and 3, 7, 10 and 14 days following single dose
  To determine inter-subject variability in intracellular dATP in cervical, vaginal, and rectal tissues and ratios of TFVdp:dATP.

OTHER OUTCOMES:
Cervicovaginal Fluid (CVF) Concentration | At 1, 3, 6, 12, 24 hours and 3, 7, 10, and 14 days following single dose.
  To determine if TFV and TAF concentration in CVF changes in proportion to TFV, TAF, and TFV-DP concentration in cervical and vaginal tissue

CONTACTS AND LOCATIONS:
Overall Officials: Angela DM Kashuba, PharmD, Principal Investigator — UNC Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Cottrell ML, Garrett KL, Prince HMA, Sykes C, Schauer A, Emerson CW, Peery A, Rooney JF, McCallister S, Gay C, Kashuba ADM. Single-dose pharmacokinetics of tenofovir alafenamide and its active metabolite in the mucosal tissues. J Antimicrob Chemother. 2017 Jun 1;72(6):1731-1740. doi: 10.1093/jac/dkx064. PMID 28369415